CLINICAL TRIAL: NCT04626219
Title: Neurobiology of Anorexia and Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Walter Kaye, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 080019
Record Dates: First submitted 2009-02-23; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Period of 12 hours where participants eat regulated meals
  Interventions: Other: Imaging; Behavioral: regulated meals
- 2 (Experimental): Period of 12 hours where participants do not eat anything
  Interventions: Other: Imaging; Behavioral: fast

INTERVENTIONS:
Other: Imaging — Imaging - Magnetic Resonance Imaging (MRI) scan of their heads
Behavioral: fast — hungry state - refrain from eating after lunch at 12 noon until 9 a.m. the next morning
  Arms: 2
Behavioral: regulated meals — standardized diet from noon until 9 a.m. the next day
  Arms: 1

SUMMARY:
The purpose of this study is to investigate areas of the brain responsible for appetite regulation. More specifically, the investigators would like to study changes in brain activation, e.g., changes in blood flow and oxygen use of the brain, during two different states: Once when the participants are hungry, and once when the participants are not hungry. The aim is to find out more about the neurobiology of Anorexia and Bulimia Nervosa by comparing women who never had an eating disorder with women who have recovered from Anorexia or Bulimia Nervosa.

DETAILED DESCRIPTION:
The main goal of this study is to explore the effects of hunger and satiety on regions in our brain in order to better understand the pathophysiology underlying restricted eating in anorexics, and overeating in women with Bulimia Nervosa. The investigators will adopt a paradigm that will model, in the laboratory, the naturalistic extremes of dietary intake practiced by women recovered from Anorexia or Bulimia Nervosa by comparing a hungry state (21-hour fast) to a satiated state (21-hour when fed). They may share an inability to precisely modulate emotionality and reward in response to salient stimuli, such as food. However, they may differ in terms of function of other pathways.

The incentive motivational drive to seek and consume food is a complex process, deriving from interrelated psychobiological factors including food's rewarding properties, an individual's homeostatic needs and cognitive ability to favor alternative behaviors. In order to examine how these factors may contribute to dysregulated feeding behavior in women recovered from Anorexia or Bulimia Nervosa, the investigators will explore measures of 1) anxiety; 2) cognitive inhibition and dysinhibition; and 3) reward.

Subjects will also be asked to undergo a Magnetic Resonance Imaging (MRI) scan of their head. This scan uses powerful magnetic fields. The magnetic fields temporarily magnetize some of the chemicals in our brain and this allows a scanner and a computer to take a very detailed picture of the structure of our brain. During the MRI, the participants will be asked to lie quietly inside the center of a large, doughnut shaped magnet for approximately 30 minutes. The participant's head will be placed in a special, helmet-like "head-holder" to help them to keep their head still. This part of the study will take place on the same day prior to the first PET scan. In this protocol, only one MRI will be done. In subjects with a questionable history of metallic fragments, an x-ray of the suspected body area will be performed before the MRI to make sure the participants have no metal fragments in their body.

In addition to fMRI scanning there are a few other tests that will be administered. This includes a Pre Study Taste Test, in order to prepare them for the fMRI taste task. Participants will be presented five solutions of sucrose (2, 4, 8, 16 and 32 weight by volume) and will then be asked to rate the pleasantness of each solution using a standard seven-point preference scale (i.e., 1=extremely dislike; 7= extremely like). They will also rate perceived sweetness of each solution using a seven-point category scale (i.e., 1=absent; 7=extreme). In addition, they will be presented variants of a tasteless solution Study participants will be asked to choose the solution that has the least taste and this solution will then be used during fMRI scanning.

The study takes place over the span of 4 consecutive days on location at the General Clinical Research Center (GCRC) at the University of California in San Diego. During day 1 of the study, lab work would be completed in the morning and several computerized and paper and pencil tasks in the afternoon. Starting at noon of Day 2 and Day 3 of the study, subject participants will undergo two identical 21-hour cycles. In one cycle, study participants will refrain from eating after lunch at 12 noon until 9 a.m. the next morning and they will engage in fMRI studies from 9 to 10:30 a.m. In the other cycle they will be given a standardized diet from noon until 9 a.m. the next day and engage in fMRI studies from 9 to10:30 a.m. The sequence of the two cycles will be randomized across subjects. Caloric consumption will also be regulated. All subjects will receive exactly the same menu over the 4 days of the study. They will eat only when at the GCRC and only when monitored by the GCRC staff. The total daily energy requirement will be calculated as 30 kcal/kg body weight per day with a 53% carbohydrate, 32% fat, 15% protein diet. Water will be provided with the amount consumed recorded. Subjects will be allowed to consume their usual amounts of caffeinated beverages but not allowed to use artificial or natural sweeteners or cream.

ELIGIBILITY:
Inclusion Criteria:

* Must have had a DSM-IV diagnosis of anorexia or bulimia nervosa
* The onset of their illness must have been at least 4 years prior to participating in this study
* Must have recovered for 12 months or more prior to entering the study.

Exclusion Criteria:

* Met diagnosis of alcohol or drug abuse or dependence in the 3 months prior to the study.
* Current diagnosis of a severe major affective or anxiety disorder or presence of other psychopathology that might interfere with ability to participate in the study.
* Organic brain syndromes, dementia, psychotic disorders or mental retardation
* Neurological or medical disorders
* Use of psychoactive medication in the 3 months prior to the study.
* Pregnancy or lactation, lack of effective birth control during 15 days before the scans.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Anterior insula (AI) and orbital frontal cortex (OFC) response to sucrose(relative to ionic water) | 5 years
  fMRI BOLD response

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kaye, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD General Clinical Research Center, San Diego, California, United States

REFERENCES:
- See also: Related Info — http://eatingdisorders.ucsd.edu